CLINICAL TRIAL: NCT06053684
Title: Comparison of Conventional Non-Invasive Ventilation and Neurally-Adjusted Ventilatory Assistance (NAVA) Non-Invasive Ventilation for the Treatment of Bronchiolitis
Brief Title: Non-Invasive Ventilation Versus Neurally-Adjusted Ventilatory Assistance (NAVA) for the Treatment of Bronchiolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-14633
Record Dates: First submitted 2023-09-06; First posted 2023-09-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Non-Invasive Mechanical Servo Ventilation Arm (Active Comparator): This arm will utilize a standard mode of non-invasive ventilation within protocol parameters.
  Interventions: Device: Standard Non-Invasive Mechanical Servo Ventilation
- Neurally-Adjusted Ventilatory Assistance (NAVA) Non-Invasive Mechanical Servo Ventilation Arm (Experimental): This arm with utilize a NAVA mode of non-invasive ventilation within protocol parameters.
  Interventions: Device: Neurally-Adjusted Ventilatory Assistance (NAVA) Non-Invasive Mechanical Servo Ventilation

INTERVENTIONS:
Device: Standard Non-Invasive Mechanical Servo Ventilation — The active comparator arm will utilize a standard non-invasive mode to provide ventilation support
  Arms: Standard Non-Invasive Mechanical Servo Ventilation Arm
Device: Neurally-Adjusted Ventilatory Assistance (NAVA) Non-Invasive Mechanical Servo Ventilation — The experimental arm will utilize a NAVA mode to provide non-invasive ventilation support
  Arms: Neurally-Adjusted Ventilatory Assistance (NAVA) Non-Invasive Mechanical Servo Ventilation Arm

SUMMARY:
This project aims to answer whether the use of a Neurally-Adjusted Ventilatory Assistance mode for non-invasive ventilation in pediatric patients with bronchiolitis results in improved comfort and reduced escalations in therapy (including intubation) when compared to using a standard mode of non-invasive ventilation. Neurally-Adjusted Ventilatory Assistance (NAVA) has been shown to result in greater synchrony then the standard mode of non-invasive ventilation. The study team hypothesizes that this improved synchrony can result in important clinical improvements when NAVA is used to treat children with bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis is a common diagnosis in pediatric hospitals and critical care units. Viral infection in younger patients often results in increased work of breathing, hypoxemia, impaired ventilation, and increased secretion burden. In some cases, treatment of severe respiratory failure includes intubation and mechanical ventilation. Current practice for patients with bronchiolitis who require hospital admission is to initially provide non-invasive ventilation to improve the patient's respiratory mechanics. This non-invasive respiratory support can range from simple nasal cannula, to high-flow nasal cannula, to non-invasive positive pressure ventilation.

The high-flow nasal cannula (HFNC) provides warm, humidified, oxygen-enriched air. Therapy commonly is prescribed with a prescribed fraction of inhaled oxygen (FiO2) delivered at 1-2 L/kg/min. This helps to improve oxygenation as the high rate of flow can "wash-out" carbon dioxide in the upper airways and thus reduce the volume of dead space ventilation.

Non-invasive ventilation (NIV) essentially provides a similar method of support as invasive ventilation without the use of endotracheal tube. Prescribed airway support is instead delivered non-invasively through a specialized nasal cannula or for larger children an occlusive facemask of appropriate size. The ventilator provides positive-end expiratory pressure (PEEP) with a prescribed delivery rate of a set inspiratory pressure (positive inspiratory pressure, or pressure control). This ventilator support enables the delivery of a set FiO2, helps maintain open airways to reduce atelectasis and allow for improved oxygenation with better V/Q matching, and improves work of breathing. The ventilator analyzes the flow generated by the patient's inspiratory effort and attempts to provide the prescribed positive inspiratory pressure at the time of the patient's own effort.

One of the major drawbacks of non-invasive ventilation for young pediatric patients with bronchiolitis is the difficulty in achieving synchrony between patient effort and ventilator-delivered positive inspiratory pressure. This is secondary to the large air leak given the non-invasive apparatus and the low inspiratory flows generated by this patient population. Thus, the ventilator and patient are often dyssynchronous which may actually increase work of breathing and agitation while impeding on the ventilatory support provided.

Neurally-Adjusted Ventilatory Assistance (NAVA) attempts to mitigate the harms of ventilator/patient dyssynchrony. This modality utilizes a specialized catheter placed into the esophagus, often via a nasogastric route, which has the capability of monitoring the electrical activity of the patient's diaphragm. This catheter can also be utilized to deliver feeds similarly to a basic nasogastric tube. The NAVA catheter monitors both the activation of the patient's diaphragm (indicating patient respiratory effort) and the strength of this activation in, referred to as the electrical activity of the diaphragm (Edi) and measured in millivolts (µV). Both human and animal studies have positively correlated the peak Edi values with work-of-breathing and demonstrated higher Edi values when respiratory pathology is present . Based on the Edi tracing, the ventilator can then deliver positive inspiratory pressure that is synchronous with both the patient's respiratory effort and proportional to the strength of this effort through a multiplier referred to as the NAVA level on the ventilator. This modality has been shown to improve patient agitation levels, reduce the need for sedating medications, and enhance synchrony in non-invasive ventilation modes.

The current practice model of the investigators entails that patients with bronchiolitis who require more than 1.5 L/kg of HFNC or require non-invasive ventilation, whether via a conventional or NAVA modality, are managed in the Pediatric Intensive Care Unit (PICU). Both modalities for non-invasive ventilation (conventional and NAVA) are used routinely. Patient respiratory status is aggregated into a value known as the Respiratory Severity Score (RSS) which accounts for respiratory rate, dyspnea, retractions, and auscultatory findings adjusted for the age of the patient. The RSS value is a validated assessment tool with good interobserver reliability between Medical Doctors (MDs), Registered Nurses (RNs), and Respiratory Therapists (RTs). It is calculated on a 4-hour basis for all patients with bronchiolitis in the investigator's PICU and helps determine clinical improvement or deterioration and better guide decisions to increase or decrease support.

While multiple physiologic studies demonstrate a reduced work of breathing with invasive NAVA ventilation, the majority of pediatric studies focused on non-invasive NAVA ventilation were designed to determine improvements in patient/ventilator synchronization. The investigators' project aims are two-fold. The study team hypothesizes that Edi levels and RSS scores will positively correlate for patients with bronchiolitis, allowing for another metric to gauge clinical status. The investigators also hypothesizes that the improved synchronization on NAVA-NIV may improve respiratory status as measured by RSS scores and Edi levels, reduce further escalations in respiratory support, shorten the length of non-invasive ventilation required, and reduce intubation rates. This improvement will be more substantial when transitioning from HFNC to NAVA-NIV compared to transitioning to conventional-NIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of two years old with a diagnosis of bronchiolitis presenting to the pediatric ICU
* Patient's provider believes there is equipoise between the use of NAVA or conventional non-invasive ventilation for the patient

Exclusion Criteria:

* Patients unable to utilize a nasogastric tube
* Patients with a diagnosis of chronic lung disease, cyanotic heart lesions, or congestive heart failure
* Patients with hypotonia
* Patients likely to require imminent intubation: >0.60 Fraction of Inspired Oxygen (FiO2); Carbon Dioxide (CO2) > 60, frequent apneas, clinician determines patient unlikely to tolerate non-invasive modality)
* Patients with hemodynamic instability, defined as the need for vasoactive medication

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Baseline Respiratory Severity Score (RSS) | Approximately one hour after Edi catheter placement
  RSS is a validated measure of severity in children with bronchiolitis, scored from 0-12 with higher numbers indicating greater severity. If able, baseline scores will be taken before randomization to either treatment arm.
Average Respiratory Severity Score (RSS) | 48 hour average, values collected at ~4 hour intervals.
  RSS is a validated measure of severity in children with bronchiolitis, scored from 0-12 with higher numbers indicating greater severity. Average RSS values over a 48-hour period will be reported for each treatment arm.
Baseline Electrical Activity of the Diaphragm (Edi) | Approximately one hour after Edi catheter placement
  Measure, in microvolts, recorded by the Edi catheter to reflect activity of diaphragmatic activation. Higher values correspond with increased diaphragmatic activation. If able, will be collected prior to randomization to either treatment arm.
Average Baseline Electrical Activity of the Diaphragm (Edi) | 48 hour average, values collected at ~4 hour intervals.
  Measure, in microvolts, recorded by the Edi catheter to reflect activity of diaphragmatic activation. Higher values correspond with increased diaphragmatic activation. Average Edi values over a 48-hour period will be reported for each treatment arm.

SECONDARY OUTCOMES:
Duration of Non-Invasive Ventilation | Time of randomization or start of non-invasive ventilation (whichever occurs last) up to 4 weeks later or time of intubation (whichever occurs first)
  The duration, in hours, that a patient requires non-invasive ventilation.
Number of participants requiring intubation | Following start of non-invasive ventilation or randomization (whichever comes last) up to 4 weeks later
  If a patient requires intubation due to bronchiolitis, this information will be recorded
Frequency of increasing ventilatory support | From hours 4-48 of the intervention period
  The number of times that a physician increases respiratory support settings on the ventilator (other than FiO2) while remaining within protocol parameters will be documented. The number of events, limited to one event per hour, of increase in respiratory support will be counted during the study period. A greater number of increases in ventilatory support will indicate inadequate response to the treatment arm intervention.
Number of patients requiring dexmedetomidine | Through 48 hour study intervention period
  The number of patients requiring dexmedetomidine will be tabulated. The use of dexmedetomidine use likely reflects patient agitation and inability to ventilate adequately on non-invasive ventilation. The use of dexmedetomidine may indicate more agitation present within a given treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Weingarten, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lodeserto FJ, Lettich TM, Rezaie SR. High-flow Nasal Cannula: Mechanisms of Action and Adult and Pediatric Indications. Cureus. 2018 Nov 26;10(11):e3639. doi: 10.7759/cureus.3639. PMID 30740281
- [Background] Javouhey E, Barats A, Richard N, Stamm D, Floret D. Non-invasive ventilation as primary ventilatory support for infants with severe bronchiolitis. Intensive Care Med. 2008 Sep;34(9):1608-14. doi: 10.1007/s00134-008-1150-4. Epub 2008 May 24. PMID 18500424
- [Background] Morley SL. Non-invasive ventilation in paediatric critical care. Paediatr Respir Rev. 2016 Sep;20:24-31. doi: 10.1016/j.prrv.2016.03.001. Epub 2016 Mar 14. PMID 27118355
- [Background] Jones ML, Bai S, Thurman TL, Holt SJ, Heulitt MJ, Courtney SE. Comparison of Work of Breathing Between Noninvasive Ventilation and Neurally Adjusted Ventilatory Assist in a Healthy and a Lung-Injured Piglet Model. Respir Care. 2018 Dec;63(12):1478-1484. doi: 10.4187/respcare.06192. Epub 2018 Sep 25. PMID 30254048
- [Background] Pham TM, O'Malley L, Mayfield S, Martin S, Schibler A. The effect of high flow nasal cannula therapy on the work of breathing in infants with bronchiolitis. Pediatr Pulmonol. 2015 Jul;50(7):713-20. doi: 10.1002/ppul.23060. Epub 2014 May 21. PMID 24846750
- [Background] Alander M, Peltoniemi O, Pokka T, Kontiokari T. Comparison of pressure-, flow-, and NAVA-triggering in pediatric and neonatal ventilatory care. Pediatr Pulmonol. 2012 Jan;47(1):76-83. doi: 10.1002/ppul.21519. Epub 2011 Aug 9. PMID 21830318
- [Background] Kallio M, Peltoniemi O, Anttila E, Pokka T, Kontiokari T. Neurally adjusted ventilatory assist (NAVA) in pediatric intensive care--a randomized controlled trial. Pediatr Pulmonol. 2015 Jan;50(1):55-62. doi: 10.1002/ppul.22995. Epub 2014 Jan 31. PMID 24482284
- [Background] Ducharme-Crevier L, Beck J, Essouri S, Jouvet P, Emeriaud G. Neurally adjusted ventilatory assist (NAVA) allows patient-ventilator synchrony during pediatric noninvasive ventilation: a crossover physiological study. Crit Care. 2015 Feb 17;19(1):44. doi: 10.1186/s13054-015-0770-7. PMID 25886793
- [Background] Liu LL, Gallaher MM, Davis RL, Rutter CM, Lewis TC, Marcuse EK. Use of a respiratory clinical score among different providers. Pediatr Pulmonol. 2004 Mar;37(3):243-8. doi: 10.1002/ppul.10425. PMID 14966818
- [Background] Duyndam A, Bol BS, Kroon A, Tibboel D, Ista E. Neurally adjusted ventilatory assist: assessing the comfort and feasibility of use in neonates and children. Nurs Crit Care. 2013 Mar-Apr;18(2):86-92. doi: 10.1111/j.1478-5153.2012.00541.x. Epub 2012 Nov 22. PMID 23419184
- [Background] Stein H, Hall R, Davis K, White DB. Electrical activity of the diaphragm (Edi) values and Edi catheter placement in non-ventilated preterm neonates. J Perinatol. 2013 Sep;33(9):707-11. doi: 10.1038/jp.2013.45. Epub 2013 May 2. PMID 23636099
- [Background] Beck J, Emeriaud G, Liu Y, Sinderby C. Neurally-adjusted ventilatory assist (NAVA) in children: a systematic review. Minerva Anestesiol. 2016 Aug;82(8):874-83. Epub 2015 Sep 16. PMID 26375790
- [Background] Vignaux L, Grazioli S, Piquilloud L, Bochaton N, Karam O, Levy-Jamet Y, Jaecklin T, Tourneux P, Jolliet P, Rimensberger PC. Patient-ventilator asynchrony during noninvasive pressure support ventilation and neurally adjusted ventilatory assist in infants and children. Pediatr Crit Care Med. 2013 Oct;14(8):e357-64. doi: 10.1097/PCC.0b013e3182917922. PMID 23863816